CLINICAL TRIAL: NCT05716932
Title: Validity of Focal Laser Photocoagulation Followed by a Single Intravitreal Ranibizumab Injection for Retinal Artery Macroaneurysm.
Brief Title: Focal Laser Single Intravitreal Ranibizumab Retinal Artery Macroaneurysm.
Acronym: RAM
Status: Completed | Type: Observational
Sponsor: Dar El Oyoun Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Wael Ahmed Ewais, Dr Wael Ewais, Dar El Oyoun Hospital
Other Study IDs: N-122-2022
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Retinal Artery Macroaneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Dual focal laser and intravitreal Ranibizumab injection — Direct and perilesional focal laser followed by a single intravitreal 0.5 mg ranibizumab (Lucentis, Genentech, Inc., South San Francisco, CA, USA) injection
  Other Names: DFL and IVR

SUMMARY:
Treatment options for Retinal artery Macroaneurysm (RAM) include focal laser photocoagulation, intravitreal anti-Vascular Endothelial Growth Factor (anti-VEGF) injection, combined anti VEGF - laser therapy, YAG hyaloidotomy and pars plana vitrectomy. Focal laser photocoagulation is applied directly to the macroaneurysm (direct lesional), its surrounding area (indirect perilesional) or a combination of both. [3-5] Anti-VEGF agents including bevacizumab and ranibizumab reduce leakage from the macroaneurysm. [3-15] YAG hyaloidotomy is used for fresh premacular hemorrhage. [16] Pars plana vitrectomy is reserved for RAM complicated by vitreous and/or premacular hemorrhage. [17]

However, there is no consensus about laser and anti VEGF treatments. Some authors use perilesional laser, while others use direct laser only. There is also no clear protocol for anti VEGF injections. Some authors report using focal laser only if multiple anti VEGF injections do not result in marked improvement. [3-17]

.

DETAILED DESCRIPTION:
Retinal arterial macroaneurysm (RAM) is an acquired localized arterial dilatation, which often occurs at second or third branches of the central retinal artery. Mostly, elderly hypertensive females above 60 years are affected. One in 4500 people over the age of 40 years is liable to develop a RAM. It may be associated with retinal vein occlusion. [1]

The natural history of a RAM can be divided into a growing phase, followed by gradual fibrosis and/ or thrombosis (closure), and then involution. A growing macroaneurysm may leak, resulting in intraretinal exudation and macular edema. It may rupture producing subretinal, intraretinal, preretinal, and / or vitreous hemorrhage. Approximately 8%-25% of RAMs undergo spontaneous involution without treatment. However, treatment is required for leaking macroaneurysms to prevent macular structural damage. [2,3]

Treatment options for RAM include focal laser photocoagulation, intravitreal anti-Vascular Endothelial Growth Factor (anti-VEGF) injection, combined anti VEGF - laser therapy, YAG hyaloidotomy and pars plana vitrectomy. Focal laser photocoagulation is applied directly to the macroaneurysm (direct lesional), its surrounding area (indirect perilesional) or a combination of both. [3-5] Anti-VEGF agents including bevacizumab and ranibizumab reduce leakage from the macroaneurysm. [3-15] YAG hyaloidotomy is used for fresh premacular hemorrhage. [16] Pars plana vitrectomy is reserved for RAM complicated by vitreous and/or premacular hemorrhage. [17]

However, there is no consensus about laser and anti VEGF treatments. Some authors use perilesional laser, while others use direct laser only. There is also no clear protocol for anti VEGF injections. Some authors report using focal laser only if multiple anti VEGF injections do not result in marked improvement. [3-17]

.

ELIGIBILITY:
Inclusion Criteria:

* We will enroll cases of RAM that had been treated by Direct and perilesional focal laser, followed by a single intravitreal ranibizumab injection a few days later, and had been followed up for at least 6 months

Exclusion Criteria:

* • RAM treated by a single approach (laser or intravitreal injections),

  * RAM treated by other anti-VEGF injections (not ranibizumab),
  * RAM with a shorter than 6 months of follow-up after combined laser and ranibizumab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective review of records of eyes with RAM; treated between February 2012 and November 2020; will be done, to collect and analyze the following data: Treatment details, features of RAM, associated retinal disease, best-corrected visual acuity (BCVA), central macular thickness (CMT), signs of RAM involution, and possible complications
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
change in best corrected visual acuity (BCVA) | 6 months
  NCVA change between baseline and final follow up at 6 months

SECONDARY OUTCOMES:
change in central macular thickness (CMT) | (Time frame: 6 months)
  between baseline and final follow up at 6 months
incidence of complications due to laser or intravitreal injection. | 6 months
  presence or absence of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy faculty of medicine, Cairo, Egypt